CLINICAL TRIAL: NCT06174792
Title: Evaluation of the Efficacy and Safety of Drospirenone in the Treatment of Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Other Study IDs: DROS_Adenomyosis
Record Dates: First submitted 2023-11-18; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; Drospirenone; progestin
MeSH Terms: conditions — Adenomyosis | interventions — drospirenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Drospirenone 4 MG — Patients who met all inclusion criteria and had no exclusion criteria would receive one tablet of Drospirenone 4mg daily for 20 weeks, starting from day 2 to day 5 of their menstrual cycle.

SUMMARY:
Adenomyosis is a common benign condition of fertile women and is characterized by dysmenorrhea, hypermenorrhea, abnormal uterine bleeding, infertility and chronic pelvic pain.

To date, no clear guidelines are available regarding the treatment of adenomyosis, however, resembling endometriosis, as it too is a sex hormone-dependent inflammatory condition, numerous hormonal and non-hormonal treatments are currently being used off-label in the treatment of this condition, succeeding in controlling, sometimes not fully efficiently, the resulting symptoms.

Among hormonal treatments, progestins have been proposed. Decreased expression of progesterone receptors (PR) A and B has been observed in adenomyotic tissue, similar to endometriosis. Progesterone induces antiproliferative activity through binding to its receptors. The observed reduction in PR expression could partially explain the pathogenesis of adenomyosis and the poor response to progestins.

Although adenomyotic tissue has lower levels of PR, a good response to high-dose topical progesterone has been demonstrated. Although several molecules have been tested, such as levonorgestrel, dienogest, and danazol, to date there are no randomized controlled trials on the use of progestins in the treatment of adenomyosis that would allow clear guidelines on their use in this setting.

Among the progestins commercially available today is drospirenone, which is used clinically as a progestin in oral contraceptives. Drospirenone is a synthetic progestin similar to human progesterone and is a potent inhibitor of mineralocorticoid activity. Drospirenone has been shown to significantly reduce the diameter and maximal volume of ovarian endometrioma, reduce dysmenorrhea, reduce postoperative anatomic and symptomatic recurrence rates, and decrease serum CA125 levels. Drospirenone also acts on the endometrium, reducing its proliferation and thus improving menorrhagia symptoms and has also been shown to reduce Ki-67 expression in the human endometrium when administered orally with and without E2.

Despite reports of these clinical effects on endometriosis, the direct effects of drospirenone on adenomyosis have never been tested.

The aim of study is to evaluate the efficacy and safety of drospirenone in the treatment of adenomyosis, and its impact on improved quality of life and sexual life.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* regular menstrual cycle;
* adenomyosis diagnosed by imaging analysis (magnetic resonance imaging [MRI] or transvaginal ultrasound);
* no other treatment for adenomyosis for at least 3 months before drospirenone administration;
* painful symptoms (lower abdominal and/or lower back pain) with a score of three points or more on the verbal pain rating scale developed by Harada et al. during the menstrual cycle.

Exclusion Criteria:

* endometriosis or uterine leiomyoma diagnosed by imaging analysis (MRI or transvaginal ultrasound);
* benign ovarian cyst including endometrioma;
* other endocrine diseases;
* severe anemia (hemoglobin concentrations <8.0 g/dL).

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Women affected by adenomyosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
reduction of the level of chronic pain assessed with Visual Analogue Scale | 20 weeks
  reduction of the level of chronic pain associated with adenomyosis

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Etrusco, Palermo, Italy